CLINICAL TRIAL: NCT04300452
Title: Carbetocin Versus Ergometrin in the Prevention of Postpartum Hemorrhage in Parturients Undergoing Caesarian Section Under Regional Anaesthesia. A Single Blind Randomized Control Trial
Brief Title: Carbetocin Versus Ergometrin in the Prevention of Postpartum Hemorrhage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Christos Koliafas, Consultant anaesthesiologist at "Elena Venizelou Hospital", National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: carbetocin-ergometrin
Record Dates: First submitted 2018-04-30; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Postpartum Hemorrhage
Keywords: carbetocin; ergometrin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Ergonovine

STUDY DESIGN:
Intervention Model Description: The parturients will be divided in two groups: the group to which carbetocin will be administered and the group to which ergometrin will be used as the main uterotonic drug. Randomization will be achieved with the help of a computer and the method ¨sealed envelope¨. In this method the investigator receives a sealed envelope either by mail or by computer, in which a random number will be placed. This number will correspond to one of the treatments. For greater relialibility in the results some exclusion criteria will be set.
Who Masked: Participant, Care Provider
Masking Description: The participants will be unaware of the treatment they will receive as well as the care provider responsible for its administration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbetocin group (Active Comparator): In the carbetocin group will be administered 100 mcg of carbetocin diluted in 100 cc of N/S 0.9% in a continuous rapid-flow intravenous infusion.
  Interventions: Drug: Carbetocin
- Ergometrin group (Active Comparator): In the ergometrine maleate group will be administered intravenously 0.2 mg of the substance slowly in a bolus administration.
  Interventions: Drug: Ergometrine Maleate

INTERVENTIONS:
Drug: Carbetocin — Administration of Carbetocin after placental detachment
  Other Names: Pabal
  Arms: Carbetocin group
Drug: Ergometrine Maleate — Administration of ergometrin after placental detachment
  Other Names: Mitrotan
  Arms: Ergometrin group

SUMMARY:
In the present study will be compared Carbetocin with ergometrin in the prevention of postpartum haemorrhage (PPH) in parturients that are undergoing caesarean section and are not presenting risk factors for PPH. As indicators will be used intraoperative blood loss, as well as the value of hemoglobin and hematocrit 24 hours after the caesarian section.

DETAILED DESCRIPTION:
In the particular study the investigators will compare the effect of Carbetocin and ergometrin in the prevention of postpartum haemorrhage. It is a prospective comparative single blind randomized study which will be carried out in the G.N.M.A. "Elena Venizelou". The protocol will be filed in an international database before the initiation of the study (eg. ClinicalTrials.gov). The sample will be constituted by parturients that will undergo Caesarean section. The parturients will be divided in two groups: the group to which carbetocin will be administered and the group to which ergometrin will be used as the main uterotonic drug. Randomization will be achieved with the help of a computer and the method ¨sealed envelope¨. In this method the investigator receives a sealed envelope either by mail or by computer, in which a random number will be placed. This number will correspond to one of the treatments. For greater reliability in the results some exclusion criteria will be set.

A consent form will be given to the parturients that will have to sign after it is explained to them the purpose of the study and that there is a rescue treatment in case of failure of the medication is administered to them. Subsequently a complete medical background will be obtained and it will be performed the standard laboratory control which includes: a blood count, coagulation parameters, biochemical parameters and an assessment by a cardiologist.

Regional anaesthesia will then be performed (spinal, epidural or combined spinal-epidural). After the embryo exit and placental detachment in the ergometrine group will be administered intravenously 0.2 mg of the substance slowly in a bolus administration, while in the carbetocin group will be administered 100 mcg of carbetocin diluted in 100 cc of N/S 0.9% in a continuous rapid-flow intravenous infusion.

The efficacy of the uterotonic drugs will be assessed with a new hemoglobin and hematocrit count 24 hours after the end of the cesarean section, as well as by intraoperative blood loss which will be calculated by weighing gauzes and compresses after the end of the operation, by the amount of blood present in the suction unit and by the blood present in the surroundings of the operating table (9). It is obvious that if necessary rescue therapy will be administered which will consist of 15 iu of oxytocin in intravenous infusion in the ergometrin group and 0.2 mg of ergometrin in slow bolus administration in the carbetocin group, as well as 3 tb of misoprostol in both groups administered per rectum.

ELIGIBILITY:
Inclusion Criteria:

* Female gender Gestating Between 18-40 years No co-morbidity

Exclusion Criteria:

* Exclusion Criteria

  * Under age parturients
  * Parturients >40 years of age
  * Multiple pregnancies
  * Parturients with abnormal placental adhesion
  * Parturients with two or more caesarian sections in the past
  * Parturients with haematological diseases
  * Parturients that receive anticoagulation therapy for a concomitant disease
  * Parturients with severe co-morbidity
  * Refusal to sign the consent form
  * Caesarian section under general anaesthesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female of reproductive age
Enrollment: 100 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2020-06-10 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
The efficacy of the uterotonic drugs wil be assessed with a new hemoglobin in gr/dl 24 hours after completion of caesarian section | 2 years
  The efficacy of the uterotonic drugs will be assessed with a new hemoglobin in g/dl 24 hours after the end of the cesarean section, as well as by intraoperative blood loss in ml which will be calculated by weighing gauzes and compresses after the end of the operation, by the amount of blood in ml present in the suction unit and by the blood present in the surroundings of the operating table.
The efficacy of the uterotonic drugs will be assessed with a new hematocrit count measured in % percentage 24 hours after completion of caesarian section. | 2 years
  The efficace of the uterotonic drugs will be assessed with a new hematocrit count measured in % percentage 24 hours after completion of caesarian section.

CONTACTS AND LOCATIONS:
Overall Officials: Nikoleta Iakovidou, Study Director — Professor of Pediatrics NKUAthens
Locations (1):
- Hospital "Elena Venizelou", Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No